CLINICAL TRIAL: NCT06952075
Title: Single-Arm, Open, Multi-Center Phase II Clinical Trial of the Efficacy, Safety, Pharmacokinetics, and Immunogenicity of GR1803 Injection in Patients With Relapsed/Refractory Multiple Myeloma Complicated by Extramedullary Plasmacytoma
Brief Title: GR1803 Injection in Patients With RRMM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GR1803-005
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myleoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GR1803 (Experimental)
  Interventions: Drug: GR1803

INTERVENTIONS:
Drug: GR1803 — D1 given at a dose of 10ug/kg, D4 given at a dose of 30ug/kg, D8 given at a dose of 180ug/kg, followed by weekly dosing up to cycle 9, and cycle 10 and onwards, every 2 weeks, with a dosing cycle of every 4 weeks

SUMMARY:
All subjects will receive GR1803 injection until intolerable toxicity or investigator-assessed disease progression occurs (except in cases of disease progression due to discontinuation of the drug as a result of an adverse event) or until the subject has been administered the drug for 2 years or until the subject withdraws consent or until the investigator determines that the subject needs to be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* 1、ECOG score 0-2 2、≥18 years of age 3、Multiple myeloma must be Complicated by Extramedullary Plasmacytoma.

Exclusion Criteria:

* 1、Prior treatment with any BCMA-targeted therapy 2、Known active CNS involvement or exhibits clinical signs of meningeal involvement of multiple myeloma 3、Known allergies, hypersensitivity, or intolerance to the study drug (teclistamab) or its excipients 4、Plasma cell leukemia , Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or primary amyloid light-chain amyloidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 years
  Sum of the proportions of patients with proven strict complete remission (sCR), complete remission (CR), very good partial remission (VGPR) and partial remission (PR)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  Time from enrollment to tumor progression or death from any cause
AE | 2 years
  adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
Study Protocol